CLINICAL TRIAL: NCT00760851
Title: Study to Investigate the Potential of Probiotics II
Brief Title: Yogurt Study in Children 2-4 Years Old Attending Daycare
Acronym: SIPPY II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Penn State University (Other)
Responsible Party: Dr. Daniel Merenstein, M.D., Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2008-01852
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-02

CONDITIONS: Infections, Respiratory; Diarrhea
Keywords: Probiotics; Child, preschool; Child Day Care Centers; Health; Immune system
MeSH Terms: conditions — Respiratory Tract Infections; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bb-12 supplemented strawberry yogurt drink
  Interventions: Other: probiotic strain Bb-12
- 2 (Placebo Comparator): Regular strawberry yogurt drink with no Bb-12 added
  Interventions: Other: no Bb-12

INTERVENTIONS:
Other: probiotic strain Bb-12 — 10^9 CFU Bb-12 per 4 oz yogurt
  Other Names: Bifidobacterium lactis 12
  Arms: 1
Other: no Bb-12 — yogurt identical to intervention yogurt, only without Bb-12 added.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effectiveness of probiotics (popularly referred to as 'live active culture' or 'good bacteria') in preventing illnesses and consequent absences from school/daycare centers of children two to four years old that attend daycare at least 3 days per week. Two yogurt drinks will be administered, one containing a specific strain of probiotic, Bb-12. It is hypothesized that children receiving the Bb-12 drink will experience fewer illnesses and absences from daycare.

In this study, participants will be asked to:

1. Give their child 4 oz. of the test yogurt each day for 90 days
2. Keep a daily diary of their child's health
3. Collect 3 stool samples from their child at the start, middle, and end of the study
4. Speak with research personnel on a bi-weekly basis regarding their child's health
5. Ensure that their child to consume any yogurts or probiotic-containing products for 110 days of the study

ELIGIBILITY:
Inclusion Criteria:

* Child aged 2 to 4 years of age
* Child attends daycare at least 3 days per week

Exclusion Criteria:

* Caregiver does not speak English or Spanish
* Caregiver does not agree to have their child refrain from cultured dairy products (yogurt) for the 105-day duration of the study
* Caregiver does not agree to collect a stool sample from their child on Day 0, 45, and 105 of the study
* Caregiver does not have a refrigerator to store the yogurt product at home
* Child is currently receiving breast milk
* Child has an allergy or hypersensitivity to milk proteins or other dairy food components such as lactose
* Child has an allergy or hypersensitivity to strawberry or red food coloring
* Child has a chronic disease
* Child has had an infection or been sick 7 days prior to starting study
* Child has had diarrhea or constipation 7 days prior to starting study
* Child has a special diet as prescribed by a medical professional
* Child has received antibiotics, antiseptics, antifungal, corticosteroids, anti-histamines, non steroidal anti-inflammatory drugs within 7 days prior to starting the study
* Child has a congenital anomaly or birth defect that requires medical care

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To determine if consumption of a yogurt drink containing Bb-12 decreases the number of absences children have from daycare/school due to illness | 90 days

SECONDARY OUTCOMES:
Determine if the yogurt supplemented with Bb-12 results in overall improved parental satisfaction due to decreased illnesses in children attending daycare/school | 90

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Merenstein, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Department of Family Medicine, Research Division, Washington D.C., District of Columbia, United States